CLINICAL TRIAL: NCT05687058
Title: Empagliflozin in ESKD - A Feasibility Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMMC-Neph-EMPESKD-01
Record Dates: First submitted 2022-09-16; First posted 2023-01-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Kidney Failure, Chronic; Heart Failure
Keywords: empagliflozin; end-stage kidney disease; pharmacokinetics; pharmacodynamics; feasibility trial; heart failure; residual kidney function; Sodium-glucose transporter type 2 inhibitor
MeSH Terms: conditions — Kidney Failure, Chronic; Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A single-center, non-randomized, two-arm intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 25 mg thrice-weekly post-hemodialysis dosing (Experimental): All participants undergoing thrice-weekly hemodialysis (HD) on the Monday-Wednesday-Friday (MWF) schedule will be assigned to the empagliflozin 25 mg thrice-weekly post-hemodialysis dosing arm (Group I).
  Interventions: Drug: Empagliflozin 25 mg thrice-weekly post-hemodialysis dosing
- Empagliflozin 10 mg daily dosing (Experimental): Patients undergoing thrice-weekly hemodialysis (HD) on the Tuesday-Thursday-Saturday (TTS) schedule, patients on twice-weekly HD, or patients on peritoneal dialysis will receive empagliflozin 10 mg daily (Group II).
  Interventions: Drug: Empagliflozin 10 mg daily dosing

INTERVENTIONS:
Drug: Empagliflozin 25 mg thrice-weekly post-hemodialysis dosing — Participants in Group I will be asked to take empagliflozin 25 mg after each hemodialysis session at home.
  Other Names: Jardiance 25 mg thrice-weekly post-hemodialysis dosing
  Arms: Empagliflozin 25 mg thrice-weekly post-hemodialysis dosing
Drug: Empagliflozin 10 mg daily dosing — Participants assigned to Group II will be asked to take empagliflozin 10 mg each morning between 8:30 and 9:30 a.m. at home.
  Other Names: Jardiance 10 mg daily dosing
  Arms: Empagliflozin 10 mg daily dosing

SUMMARY:
The aim of this study is to learn about the safety of empagliflozin in dialysis patients as a preparation for a future large clinical trial. Empagliflozin has been approved by the Food and Drug Administration for the treatment of either type 2 diabetes, heart failure, or chronic kidney disease among patients not on dialysis. The use of empagliflozin has not been studied or approved among patients on dialysis for kidney failure because empagliflozin acts on the kidneys. However, recent experimental studies have indicated that empagliflozin may provide direct heart benefits. Some dialysis patients have substantial residual kidney function, which may be protected by empagliflozin.

Participants will be given empagliflozin for three (3) months on top of the standard of care (usual medical care for participants' condition) and will be followed up until one (1) month after the last dose. The investigators will collect information about participants' general health, obtain blood, urine, and imaging studies, check home blood pressure, monitor home blood sugar levels, and ask health-related questions to assess the safety and potential benefits of empagliflozin over four (4) months, including one month before the three (3)-month empagliflozin treatment.

DETAILED DESCRIPTION:
The incidence of end-stage kidney disease (ESKD) in the US ranks among the highest in the world. ESKD is the last phase of chronic kidney disease when the kidneys are functioning below 10-15% of normal capacity, and the patient is on dialysis. According to the US Renal Data System (USRDS), 120,834 individuals started dialysis and nearly 524,000 people were living on dialysis in 2017.1 Although advancement in technology and general medical care has led to a modest decrease in mortality among dialysis patients, their mortality rate remains extremely high at approximately 16.5 per 100 patient-years. The leading cause of death among dialysis patients is cardiovascular disease (CVD), accounting for almost 45% of deaths. Unfortunately, established therapies to prevent incident CVD in the general population, such as renin-angiotensin system inhibitors or statins, have not been shown to be effective in the dialysis population.

Sodium-glucose transporter type 2 (SGLT2) inhibitors are originally approved by FDA for the treatment for type 2 diabetes. SGLT2 is localized to the brush border of the early proximal tubule, and hence, SGLT2inhibitors induce osmotic diuresis and natriuresis but do not activate the systemic renin-angiotensin-aldosterone system.2 Recent clinical trials have consistently shown their potent renal and cardiovascular benefits in both diabetic and non-diabetic patients, which cannot be explained only by their glucose-lowering and diuretic properties. In fact, diuretics have not been shown to reduce cardiovascular mortality and such benefits of SGLT2 inhibitors are clear even among non-diabetic populations.3-5 Their renoprotective effect potentially extends to the dialysis population where residual kidney function (RKF) still plays a major role in solute clearance and volume control and has a strong association with patient outcomes.6 Patients who retain greater RKF can consume a more liberal diet and have better nutritional status, less pill burden, better blood pressure, and less interdialytic fluid gain with less frequent intradialytic hypotension, as well as greater quality of life and better survival.6 The pathophysiology underlying the cardiovascular benefits of SGLT2 inhibitors are yet to be fully elucidated, but a recent in-vitro studies indicate its direct effects on cardiomyocytes. Therefore, the investigators hypothesize that dialysis patients also benefit from SGLT2 inhibitors even if they do not have any RKF.

Efficacy and safety studies with SGLT2 inhibitors did not enroll end-stage kidney disease (ESKD) patients on dialysis. Empagliflozin, canagliflozin, and dapagliflozin can be started if the glomerular filtration rate is more than 20-25 mL/min per 1.73 m2 and can be continued until dialysis initiation or kidney transplant. From a pharmacokinetics standpoint, those SGLT2 inhibitors are extensively metabolized by glucuronidation into inactive metabolites, and are not likely to cause dose-dependent toxicity even in ESKD. Nevertheless, extra caution is necessary for their use in the setting of ESKD because SGLT2 inhibitors are not well dialyzable due to large distribution volumes and high protein binding rates.

Our overall goal is to conduct a non-randomized feasibility clinical trial of empagliflozin in the dialysis population to obtain data that will help plan future larger, sufficiently powered efficacy clinical trials. The investigators plan to enroll a total of 24 dialysis patients (18 patients on hemodialysis and 6 patients on peritoneal dialysis). After one month of the run-in period, participants will take oral empagliflozin for 3 months.

*Hemodialysis is a form of renal replacement therapy that utilizes an external filter (dialyzer) to remove wastes from the bloodstream. Peritoneal dialysis utilizes the peritoneum as a filter to remove wastes.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years;
2. diagnosis of end-stage kidney disease requiring dialysis, and
3. ability to provide informed consent.

Exclusion Criteria:

1. systolic blood pressure <100 mm Hg (pre-dialysis for HD patients)
2. two or more episodes of urinary tract infection within the last 12 months
3. history of urinary retention or urinary tract obstruction
4. liver cirrhosis
5. advanced heart failure requiring heart assist device or inotropic support
6. heart or liver transplant recipient
7. major surgery performed within the last 3 months ("major" per the investigator's assessment)
8. major surgery scheduled within 3 months after screening ("major" per the investigator's assessment)
9. active cancer
10. pregnant or lactating women
11. known allergy or hypersensitivity to any SGLT2 inhibitors
12. history of ketoacidosis during the last 12 months
13. any other medical condition considered unappropriated by their nephrologists or a study physician (i.e., cachexia, short life expectancy, or uncontrolled personality/phycological disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible patients out of screened patients | During the screening process
Success rate of obtaining consent from those eligible patients | During the enrollment process
Proportion of missing doses | 3 months
  The investigators will do pill count using medication bottles and calculate the proportion of missing doses from each patient.
Proportion of empagliflozin discontinuation | 3 months
  Proportion of participants who discontinue empagliflozin for any reason
Dropout rate | 3 months
  Proportion of participants who dropped out from the study for any reason
Length of time on continuous glucose monitoring | 3 months
  Continuous glucose monitoring will be done for up to 14 days.
Completion rate of timed urine collection | 3 months
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | Immediately before the first dose
  The 1st blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 30 minutes of the first dose
  The 2nd blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 1 hour of the first dose
  The 3rd blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 1.5 hours of the first dose
  The 4th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 2 hours of the first dose
  The 5th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 3 hours of the first dose
  The 6th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 4 hours of the first dose
  The 7th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 8 hours of the first dose
  The 8th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 12 hours of the first dose
  The 9th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Blood empagliflozin concentrations after the first dose among patients on peritoneal dialysis | At 24 hours of the first dose
  The 10th blood draw for the pharmacokinetic study among patients on peritoneal dialysis
Random blood empagliflozin level | At Month 1
  Time since the last dose will be recorded.
Random blood empagliflozin level | At Month 2
  Time since the last dose will be recorded.
Random blood empagliflozin level | At Month 3
  Time since the last dose will be recorded.
Peritoneal dialysis clearance of empagliflozin | At Month 3
  Peritoneal dialysis fluid will be collected for 24 hours.

SECONDARY OUTCOMES:
Number of Participants with Hepatic injury | 3 months
  defined by an elevation of AST and/or ALT >3-fold upper limit of normal (ULN) combined with an elevation of total bilirubin >2-fold ULN measured, and/or marked peak aminotransferase (ALT and/or AST) elevations ≥5-fold ULN
Number of Participants with Ketoacidosis | 3 months
  defined by elevated serum beta hydroxybutyrate ≥3.0 mmol/L
Number of Participants with Lower limb amputation | 3 months
  defined by any non-trauma-related event leading to a lower limb procedure of amputation, auto-amputation or disarticulation
Number of Participants with Symptomatic urinary tract infection | 3 months
  defined by symptoms consistent with urinary tract infection plus pyuria and bacteriuria - urine culture sample has to be taken and sent to central lab for confirmation of the diagnosis
Number of Participants with genital infection | 3 months
  per patient report
Number of Participants with Tinea cruris | 3 months
  per patient report
Number of Participants with Nausea | 3 months
  per patient report
Number of Participants with Vomiting | 3 months
  per patient report
Number of Participants with Skin and soft tissue infection | 3 months
  per patient report
Days on continuous glucose monitoring (CGM) | Run in (within one month prior to the study start)
  Per CGM report
Days on continuous glucose monitoring (CGM) | At Month 0
  Per CGM report
Days on continuous glucose monitoring (CGM) | At Month 2
  Per CGM report
% Time of active CGM | Run in (within one month prior to the study start)
  Per CGM report
% Time of active CGM | At Month 0
  Per CGM report
% Time of active CGM | At Month 2
  Per CGM report
Average glucose | Run in (within one month prior to the study start)
  Per CGM report
Average glucose | At Month 0
  Per CGM report
Average glucose | At Month 2
  Per CGM report
Glucose management indicator (estimated A1C level based on the average glucose level from CGM readings for 14 or more days) | Run in (within one month prior to the study start)
  Per CGM report
Glucose management indicator (estimated A1C level based on the average glucose level from CGM readings for 14 or more days) | At Month 0
  Per CGM report
Glucose management indicator (estimated A1C level based on the average glucose level from CGM readings for 14 or more days) | At Month 2
  Per CGM report
Glucose variability | Run in (within one month prior to the study start)
  Per CGM report
Glucose variability | At Month 0
  Per CGM report
Glucose variability | At Month 2
  Per CGM report
Time in very high range (%) | Run in (within one month prior to the study start)
  Percent time for plasma glucose >250 mg/dL
Time in very high range (%) | At Month 0
  Percent time for plasma glucose >250 mg/dL
Time in very high range (%) | At Month 2
  Percent time for plasma glucose >250 mg/dL
Time in high range (%) | Run in (within one month prior to the study start)
  Percent time for plasma glucose >180 to 250 mg/dL
Time in high range (%) | At Month 0
  Percent time for plasma glucose >180 to 250 mg/dL
Time in high range (%) | At Month 2
  Percent time for plasma glucose >180 to 250 mg/dL
Time in target range (%) | Run in (within one month prior to the study start)
  Percent time for plasma glucose >70 to 180 mg/dL
Time in target range (%) | At Month 0
  Percent time for plasma glucose >70 to 180 mg/dL
Time in target range (%) | At Month 2
  Percent time for plasma glucose >70 to 180 mg/dL
Time in low range (%) | Run in (within one month prior to the study start)
  Percent time for plasma glucose >54 to 70 mg/dL
Time in low range (%) | At Month 0
  Percent time for plasma glucose >54 to 70 mg/dL
Time in low range (%) | At Month 2
  Percent time for plasma glucose >54 to 70 mg/dL
Time in very low range (%) | Run in (within one month prior to the study start)
  Percent time for plasma glucose 54 mg/dL or lower
Time in very low range (%) | At Month 0
  Percent time for plasma glucose 54 mg/dL or lower
Time in very low range (%) | At Month 2
  Percent time for plasma glucose 54 mg/dL or lower
Number of Participants with Hypoglycemia levels 1 | Run in (within one month prior to the study start)
  Plasma glucose <70 mg/dL for ≥15 minutes
Number of Participants with Hypoglycemia levels 1 | At Month 0
  Plasma glucose <70 mg/dL for ≥15 minutes
Number of Participants with Hypoglycemia levels 1 | At Month 2
  Plasma glucose <70 mg/dL for ≥15 minutes
Number of Participants with Hypoglycemia levels 2 | Run in (within one month prior to the study start)
  Plasma glucose <54 mg/dL for ≥15 minutes
Number of Participants with Hypoglycemia levels 2 | At Month 0
  Plasma glucose <54 mg/dL for ≥15 minutes
Number of Participants with Hypoglycemia levels 2 | At Month 2
  Plasma glucose <54 mg/dL for ≥15 minutes
Number of Participants with Prolonged hypoglycemia | Run in (within one month prior to the study start)
  Plasma glucose <54 mg/dL for ≥2.0 hours
Number of Participants with Prolonged hypoglycemia | At Month 0
  Plasma glucose <54 mg/dL for ≥2.0 hours
Number of Participants with Prolonged hypoglycemia | At Month 2
  Plasma glucose <54 mg/dL for ≥2.0 hours
Changes from baseline to Month 3 in left ventricular end-diastolic volume | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in left ventricular end-systolic volume | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in left ventricular mass index | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in left ventricular ejection fraction | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in left ventricular diastolic function | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in longitudinal global strain | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in radial global strain | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in circumferential global strain | 3 months
  To be evaluated by transthoracic echocardiogram (optional)
Changes from baseline to Month 3 in home systolic blood pressure | 3 months
Changes from baseline to Month 3 in home diastolic blood pressure | 3 months
Changes from baseline to Month 3 in Kidney Disease Quality of Life (KDQOL)-36 questionnaire | 3 months
  Details are available at the URL below. https://www.rand.org/content/dam/rand/www/external/health/surveys_tools/kdqol/kdqol36.pdf
Changes from baseline to Month 3 in residual kidney function | 3 months
  Renal urea clearance
Changes from baseline to Month 3 in hemoglobin | 3 months
Changes from baseline to Month 3 in erythropoiesis stimulating drug dose | 3 months
Hospitalization/Emergency room visit rate for heart failure | 3 months
Cardiovascular mortality | 3 months
All-cause mortality | 3 months
Changes Estimated glomerular filtration rate (GFR) from baseline to Month 3 | 3 months
  Estimated by Cystatin C and beta-2 macroglobulin

OTHER OUTCOMES:
Semi-structured interview | 3 months
  The results would be qualitative and provide data that are needed to improve the enrollment efficiency and protocol adherence. This will be done by tracking eligible screened patients who then go on to participate in the study as well as overall participant compliance with study procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitsugu Obi, MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Jackson Medicall Mall Dialysis Clinic, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author, Dr. Yoshitsugu Obi, MD. The data are not publicly available due to restrictions e.g. their containing information that could compromise the privacy of research participants.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available upon request after one month until 60 months of the publication of the manuscript.

DOCUMENTS (1):
  • Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT05687058/ICF_000.pdf